CLINICAL TRIAL: NCT05447936
Title: Estimation of Daily Optimal Efficacy Dose (OED) of Jarlsberg Cheese in Order to Increase the Osteocalcin Level in Young, Active Norwegian Cross-country Skiers (XCS)
Brief Title: Dose Estimation of Jarlsberg Cheese in Young, Active Norwegian Cross-country Skiers (XCS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meddoc (Other)
Collaborators: Tine (Industry)
Responsible Party: Principal Investigator, Prof Stig Larsen, Professor Emeritus, Meddoc
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: XCS-Jarlsberg/IC_2021
Record Dates: First submitted 2022-06-28; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Healthy Nutrition
Keywords: Jarlsberg cheese
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: The participants were divided into men and women. Within each of these two arms, a three-step dose escalation was performed according to a Respons Surface Pathway procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Female arm (Active Comparator): Ten healthy active female XCS past the age of 18 years were included. The duration of the study was 12 weeks divided in three dose-escalation periods of four weeks. In the first 4-week period all the participants was given 47gram Jarlsberg cheese daily. Based on the change in serum Osteocalcin level, the daily intake of Jarlsberg cheese for the next 4-week periode was desided in accordance with the RSP procedure
  Interventions: Dietary Supplement: Jarlsberg cheese
- Male arm (Active Comparator): Ten healthy active male XCS past the age of 18 years were included. The duration of the study was 12 weeks divided in three dose-escalation periods of four weeks. In the first 4-week period all the participants was given 47gram Jarlsberg cheese daily. Based on the change in serum Osteocalcin level, the daily intake of Jarlsberg cheese for the next 4-week periode was desided in accordance with the RSP procedure
  Interventions: Dietary Supplement: Jarlsberg cheese

INTERVENTIONS:
Dietary Supplement: Jarlsberg cheese — Jarlsberg cheese is a regular cheese for free sale in grocery stores. The allotted amount of cheese was taken orally each day
  Other Names: Vitamin D

SUMMARY:
The main aim was to estimate the daily OED of Jarlsberg cheese related to increased total serum Osteocalcin (tOC) level in young, active female and male Cross-country skiers (XCS).

The study population consists of active Cross-country Skiers (XCS) of both genders above 18 years of age.

The optimal daily intake of Jarlsberg cheese is assumed to have a dose window of [20 - 100] gram/day and a starting dose of 47 gram/day for both female and male.

The study was performed equally as an open, two-armed within-patient Response Surface Pathway (RSP) trial with three design level and skewed starting dose.

The main response variable will be the change in the tOC level after four weeks from baseline of the given design level.

Participants, who fulfil the inclusion criteria, do not meet any of the exclusion criteria and willing to give informed consent to participate will receive an appointment for starting the study. All demographic data, social factors, history of disease and vital signs will be recorded at screening.

Blood samples was taken at screening and every four weeks. Muscle strength, Peak VO2 and BMD recorded at screening and at the end of the clinical part week12.

Ten female and 10 male XCS divided was be included, perform and completed the study.

DETAILED DESCRIPTION:
Aim

* To estimate the daily OED of Jarlsberg cheese related to increased total serum Osteocalcin (tOC) level in young, active female and male Cross-country skiers (XCS).
* To estimate the effect of daily Jarlsberg cheese intake on increased, muscle strength, peak VO2 and bone mineral density.

Study population: The study population consists of active Cross-country Skiers (XCS) of both genders above 18 years of age. The study is separated in one female and one male XCS study arm.

Trial treatment:The optimal daily intake of Jarlsberg cheese is assumed to have a dose window of [20 - 100] gram/day and a starting dose of 47 gram/day for both female and male. The cheese is received in package of 250 gram divided in 16 slices of 15.625 gram. 47 gram represents 3 slices of cheese.

Design and randomization: The female and the male arms of the study will be performed equally as an open, two-armed within-patient Response Surface Pathway (RSP) study with three design level and skewed starting dose. The two parts will be performed separately in parallel with identical RSP-design.

The main outcome variable will be categorized in the following four categories:

1. Low to moderate increase in the tOC level: [0- 10%> the last 4 weeks
2. High increase in the tOC level: ≥10% the last 4 weeks
3. Low to moderate decrease in the tOC level: <0 - 10% > the last 4 weeks
4. High decrease in the tOC level: ≥ 10% the last 4 weeks

Ten XCS in both arms will be included in the first design level and all receiving the starting dose of Jarlsberg cheese every day in four weeks. The individual increase in tOC from baseline to four weeks will be used to calculate the doses for the XCS in the second design level. The individual increase tOC in the second design will decide the daily doses of cheese to be used in the third design level.

The OED for healthy women in pre-menopausal age was previously estimated to 57-gram Jarlsberg cheese per day. It is unknown if this OED will be different from active XCS and dependent of gender and age.1 The initial dose window in this study was set to [20 - 100] gram based on the previous dose-response study in healthy pre-menopausal women.

Based on prior knowledge, the tOC follows a quadratic function in Jarlsberg cheese dose.1 The Osteocalcin seem to increase with increasing dose until a maximum (OED) and reduces for higher intake of the cheese. OED might be below the midpoint of the initial dose window of 60 gr/day. In order to optimize the estimation procedure with the skewed starting dose of 47g/day or 3 slices of Jarlsberg cheese will be chosen.

This gives an adjusted starting dose window of [20 - 74] gr/day. In case the results from all the five XCS of equal gender in the first design level reports an increase < 10% in the tOC level, the RSP-procedure recommend a maximum escalation in the daily intake of Jarlsberg cheese in the second design level. The new starting dose-window will then be change with the previously used starting dose as lower boundary.2 In the present study the adjusted dose-window for the second design level will then be [47 - 85] g/day with the new starting dose of 66 g/day. In case the results obtained at the design level recommend different doses to be used for the next level, the common RSP procedure will be followed.

Main variables: The main response variable will be the change in the tOC level after four weeks from baseline of the given design level. The osteocalcin ratio R0 defined as the ratio between carboxylated osteocalcin (uOC) and under-carboxylated osteocalcin (ucOC) = [cOC / ucOC], together with vitamin K2 and the different variants MK-7, MK-8,MK- 9 and MK-9(4H) will be used as secondary variables. Diet registration will be performed at screening and every 4 weeks. Additionally, increase in Muscle strength, Peak VO2 and Bone mineral density (BMD) will be measurement at screening and at the end of the study (week 12). Blood samples for measurements of HbA1C and Lipids; Collagen (CTX-1) and Procollagen (PINP); Estradiol and Testosterone; Progesterone and FSH will be taken at screening and at the last visit week 12 in the study. The Common Terminology Criteria for Adverse Events version 4.0 (CTCAE) will be used for registration of Adverse Events (AE) and toxicity score at every investigation visit.

Study procedure: Participants, who fulfil the inclusion criteria, do not meet any of the exclusion criteria and willing to give informed consent to participate will receive an appointment for starting the study. All demographic data, social factors, history of disease and vital signs will be recorded at screening.

Blood samples for measurements of Haematological and biochemical variables, HbA1C and Lipids; Collagen (CTX-1) and Procollagen (PINP); Estradiol and Testosterone; LH, FSH and SHBG will be taken at screening. Additionally, muscle strength, Peak VO2 and BMD will be recorded before starting the clinical part.

The design consists of three design levels within each study arm. Measurement will be taken at screening and every four weeks after daily intake of the decided dose of Jarlsberg cheese. All the participants will be asked not to change anything in their common intake of food during the study except for replacing other cheese with the received daily dose of Jarlsberg. Clinical examination, blood sampling for osteocalcin measurement and diet registration will be performed every fourth week during the study including follow-up. The physical examination includes registration of vital signs, CTCAE and change in concomitant medication. Blood sampling will be taken for measurements of tOC, cOC and ucOC and vitamin K. Blood sampling for measurements of HbA1C and Lipids; Collagen (CTX-1) and Procollagen (PINP); Estradiol and Testosterone; LH and FSH; haematological and bio-chemical variables will be taken at the last visit in the study (week 12). Additionally, muscle strength, Peak VO2 and BMD will be recorded at week 12.

Sample size: Ten female and 10 male XCS divided will be included, perform and complete the study. The minimum number of participants recommended in each arm in a within-patient RSP model is 8

ELIGIBILITY:
Inclusion Criteria:

-Healthy active XCS of both genders past the age of 18 years

Exclusion Criteria:

* Eating disorder
* Pregnancy
* Known gastrointestinal disorder
* Abnormal liver or kidney function.
* Diabetes
* Suffering from verified cancer
* Under systemic treatment with corticosteroids or other immunosuppressive drugs the last 3 weeks before start of the trial treatment.
* Participating in another clinical trial with pharmaceuticals the last six weeks before start of this trial treatment.
* Lactose intolerance or known milk product allergy
* Not able to understand information.
* Do not want or not able to give written consent to participate in the study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — self-representation of gender identity
Enrollment: 20 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
tOC | Week 0
  Total serum Osteocalcin in ng/ml
tOC | Week 4
  Total serum Osteocalcin in ng/ml
tOC | Week 8
  Total serum Osteocalcin in ng/ml
tOC | Week 12
  Total serum Osteocalcin in ng/ml

SECONDARY OUTCOMES:
K2 | Week 0
  Vitamin K2 vitamers in ng/ml
K2 | Week 4
  Vitamin K2 vitamers in ng/ml
K2 | Week 8
  Vitamin K2 vitamers in ng/ml
K2 | Week 12
  Vitamin K2 vitamers in ng/ml
BMD | Week 0
  Bone mineral density in g/cm2
BMD | Week 12
  Bone mineral in g/cm2
PINP | Week 0
  Procollagen type 1 N-terminal propeptide in ng/ml
PINP | Week 12
  Procollagen type 1 N-terminal propeptide in ng/ml
CTX | Week 0
  Serum cross-linked C-telopeptide type I collagen in ng/ml
CTX | Week 12
  Serum cross-linked C-telopeptide type I collagen in ng/ml
MS | Week 0
  Muscle strength in kg
MS | Week 12
  Muscle strength in kg

CONTACTS AND LOCATIONS:
Overall Officials: Stig E Larsen, PhD, Principal Investigator — Meddoc
Locations (1):
- Meddoc, Skjetten, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No
The data from this study will not be shared